CLINICAL TRIAL: NCT01013805
Title: A Phase II Trial of Integrated Preoperative Radiotherapy and Chemotherapy With Oxaliplatin 5-FU and Folinic Acid in Patients With Locally Advanced Rectal Cancer
Brief Title: Preoperative Radiotherapy and Chemotherapy in Patients With Locally Advanced Rectal Cancer
Acronym: PROArCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 09.01; ACTRN12610000175077 (Registry Identifier: Australia New Zealand Clinical Trials Registry)
Record Dates: First submitted 2009-10-08; First posted 2009-11-16 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Rectal Cancer
Keywords: Rectal Cancer; Chemotherapy; Radiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Integrated Preoperative Radiotherapy (external beam radiotherapy) and Chemotherapy (Oxaliplatin, Fluorouracil and Leucovorin), then surgical resection.
  Interventions: Radiation: External Beam Radiotherapy; Drug: Oxaliplatin; Drug: Fluorouracil; Drug: Leucovorin; Procedure: Surgical Resection

INTERVENTIONS:
Radiation: External Beam Radiotherapy — Weeks 3 to 5: radiotherapy 25.2 Gy in 14 fractions over 3 weeks with 85 mg/m2 oxaliplatin on the first day and continuous infusion 5-FU 200 mg/m2/day on the days of radiotherapy.
  Weeks 8-10: as per Weeks 3-5
  Other Names: Radiotherapy; RT
Drug: Oxaliplatin — Week 1: Oxaliplatin 100 mg/m2 Day 1 (over 2 hours), leucovorin 200mg/m2 Day 1 concurrent with oxaliplatin over 2 hrs (then 5-FU).
  Weeks 3 to 5: radiotherapy 25.2 Gy in 14 fractions over 3 weeks with 85 mg/m2 oxaliplatin on the first day Week 6: as per Week 1, Weeks 8-10: as per Weeks 3-5 Weeks 11: as per Week 1.
Drug: Fluorouracil — Week 1: (after Oxaliplatin and leucovorin)5-FU 400mg/m2 bolus Day 1, then 5-FU continuous infusion 2.4 g/m2 over 46 hours from Day 1.
  Weeks 3 to 5: radiotherapy 25.2 Gy in 14 fractions over 3 weeks with 85 mg/m2 oxaliplatin on the first day and continuous infusion 5-FU 200 mg/m2/day on the days of radiotherapy Week 6: as per Week 1, Weeks 8-10: as per Weeks 3-5 Weeks 11: as per Week 1.
  Leucovorin 200 mg/m2 Day 1 concurrent with Oxaliplatin over 2 hrs, then 2nd: 5-FU 400 mg/m2 bolus Day 1, then 3rd: 5-FU continuous infusion 2.4 g/m2 over 46 hours from Day 1
Drug: Leucovorin — Week 1: Oxaliplatin 100 mg/m2 Day 1 (over 2 hours), leucovorin 200mg/m2 Day 1 concurrent with oxaliplatin over 2 hrs (then 5-FU) Week 6: as per Week 1, Weeks 11: as per Week 1.
Procedure: Surgical Resection — Surgery is to be performed according to the standard procedure for locally advanced rectal cancer 4 to 6 weeks after completion of the integrated preoperative radiotherapy with FOLFOX chemotherapy regimen.

SUMMARY:
The aims of the trial are (1) to determine the tolerability rate in the setting of a multi-centre study and (2) to determine secondary tolerability endpoints, toxicity rates and complete pathologic response rate in patients with locally advanced rectal cancer who are treated with an integrated preoperative radiotherapy with FOLFOX chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated and pathologically proven adenocarcinoma of the rectum.
* MRI staged T3 or T4, any N.
* Lower border of tumour must be within 12 cm of anal verge.
* Age greater than or equal to 18 years.
* ECOG Performance Status 0-1 (Appendix 2)
* Absolute neutrophil count greater than or equal to 1.5 x 109/L, haemoglobin greater than or equal to 90 g/L, and platelets greater than or equal to 100 x 109/L.
* Adequate renal function: GFR greater than or equal to 55 mL/min (derived from serum creatinine e.g. using the Cockcroft-Gault formula or measured by radioisotopic techniques).
* Bilirubin and ALT less than or equal to 1.5 x upper limit of normal.
* No symptomatic peripheral neuropathy greater than or equal to grade 2.
* Male or non-pregnant, non-lactating female. Patients on study with reproductive potential, or female partners with reproductive potential, must use an effective contraceptive.
* Has provided written informed consent for participation in this trial

Exclusion Criteria:

* Presence of metastatic disease.
* Prior pelvic radiotherapy
* Febrile intercurrent illness or infection.
* Previous history of unstable angina
* Cardiac arrhythmia which in the opinion of the investigator would compromise the safe delivery of protocol treatment
* Acute coronary syndrome even if controlled with medication
* Myocardial infarction within the last 12 months
* Concurrent treatment with other anti-cancer therapy.
* Significant medical condition which in the opinion of the investigator would compromise the planned delivery of the chemotherapy and radiotherapy or which may be potentially exacerbated by these modalities.
* Locally recurrent rectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Tolerability Rate of patients treated with integrated pre-operative radiotherapy with FOLFOX chemotherapy regimen | End of preoperative treatment (11 weeks)

SECONDARY OUTCOMES:
Complete pathologic response rate following the completion of treatment | Determined post-surgery
Treatment Related Toxicity rates | Determined after preoperative treatment and 30 days post-surgery
Dose Intensity of the treatment drug | End of preoperative treatment (11 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Ngan, Study Chair — Trans Tasman Radiation Oncology Group
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

REFERENCES:
- See also: Click here for more information about this study on the TROG website — http://www.trog.com.au